CLINICAL TRIAL: NCT06815302
Title: TURN-IT FOG: A Novel Intervention to Improve Turning in People With PD and Freezing of Gait
Brief Title: TURN-IT FOG: Improving Turning and Freezing of Gait in People With PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Martina Mancini, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MJFF-024692; MJFF-024692 (Other Grant/Funding Number: Michael J. Fox Foundation for Parkinson's Research)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Freezing of Gait Symptoms in Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic balance exercise intervention group (Experimental): Six weeks of exercise intervention to improve gait disturbances.
  Specific participant procedures in experimental and active control interventions are simplified to preserve study blinding.
  Interventions: Behavioral: Experimental intervention
- Strength training exercise intervention group (Active Comparator): Six weeks of exercise intervention to improve gait disturbances.
  Specific participant procedures in experimental and active control interventions are simplified to preserve study blinding.
  Interventions: Behavioral: Active intervention

INTERVENTIONS:
Behavioral: Experimental intervention — Specific participant procedures in experimental and active control interventions are simplified to preserve study blinding.
  Arms: Dynamic balance exercise intervention group
Behavioral: Active intervention — Specific participant procedures in experimental and active control interventions are simplified to preserve study blinding.
  Arms: Strength training exercise intervention group

SUMMARY:
The goals of this clinical trial are to 1) learn how two different rehabilitation interventions for PD can reduce Freezing of Gait (FOG) in people with Parkinson's disease, as assessed by patients, clinicians, and wearable sensors, and 2) to explore whether two different rehabilitation intervention can reduce FOG and improve daily life mobility in people with FOG sufficiently to justify a clinical trial.

Participants will:

* Be randomly assigned to one of two intervention groups (turning-focused agility exercise or strength-based exercise)
* Have one-on-one training sessions three times per week for 6 weeks
* Perform in-lab assessments before beginning and after completing the study intervention
* Use wearable mobility sensors during daily life to measure their walking and balance

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD from movement disorders neurologist with the United Kingdom Brain Bank criteria of bradykinesia with one or more of the following - rest tremor, rigidity, and balance problems not from visual, vestibular, cerebellar or proprioceptive conditions
* reporting FOG in the New Freezing of Gait questionnaire (N-FOGQ)
* Hoehn & Yahr stages II-IV
* ages 50-80 years old
* cognitive ability sufficient to participate in testing procedures and exercise classes
* be willing and able to participate in exercise intervention 3x/week for 6 weeks

Exclusion Criteria:

* Major musculoskeletal or neurological disorders, structural brain disease, epilepsy, acute illness or health history, other than PD, significantly affecting gait and turning (i.e., musculoskeletal disorder, vestibular problem, head injury, stroke, cardiac disease)
* medical condition or medications that precludes moderate-intensity exercise
* Montreal Cognitive Assessment (MoCA) ≤21 or inability to follow directions
* excessive use of alcohol or recreational drugs
* recent change in medication
* inability to stand and walk for 2 minutes without an assistive device

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient- Perceived Freezing of Gait Severity | From enrollment/randomization through intervention; 8 weeks
  Change in freezing of gait severity with the intervention (scored in likert scale by the patient; 3 = Much improved, 2 = Somewhat improved, 1 = Minimally improved, 0 = No change, -1 = Minimally worse, -2 = Somewhat worse, -3 = Much worse)
Clinician- Perceived Freezing of Gait Severity | From enrollment/randomization through intervention; 8 weeks
  Change in freezing of gait severity with the intervention (scored in likert scale by the clinician; 3 = Much improved, 2 = Somewhat improved, 1 = Minimally improved, 0 = No change, -1 = Minimally worse, -2 = Somewhat worse, -3 = Much worse
Sensors-based Freezing of gait severity | From enrollment/randomization through intervention; 8 weeks
  Freezing of Gait Index calculated during a 360 degrees turning in place from wearable sensors; continuous scale, with a higher positive score meaning a greater level of freezing of gait.

SECONDARY OUTCOMES:
Time Spent in FOG during daily life | From enrollment/randomization through intervention; 8 weeks
  % time spent FOG compared to walking during daily life calculated from wearable sensors

CONTACTS AND LOCATIONS:
Overall Officials: Martina Mancini, PhD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - Oregon Health and Science University, Portland, Oregon
- University of São Paulo, Bauru Campus, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to study outcomes measures will be publicly shared
Time Frame: Data would be available 6 months after publication.
Access Criteria: Data will be deposited on Zenodo https://zenodo.org/records/12548174
URL: https://zenodo.org/records/12548174